CLINICAL TRIAL: NCT02154737
Title: A Phase I, Open-label, Dose Escalation Study of Gemcitabine and Pulse Dose Erlotinib in Second Line Treatment of Advanced Pancreatic Cancer
Brief Title: Gemcitabine and Pulse Dose Erlotinib in Second Line Treatment of Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tony Reid, M.D., Ph.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Tony Reid, M.D., Ph.D., Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121359
Record Dates: First submitted 2013-06-14; First posted 2014-06-03 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Gemcitabine; Gemzar; erlotinib; Tarceva
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib and gemcitabine (Experimental): Erlotinib will be administered orally on Days 2-4 and Days 16-18 of a 28-day cycle in serial cohorts with doses of 750mg, 1000mg, 1250mg, 1500mg, 1750mg, and 2000mg
  Gemcitabine will be administered intravenously at 1000 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Erlotinib

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered intravenously at 1000 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
  Other Names: Gemzar
Drug: Erlotinib — Erlotinib will be administered orally on Days 2-4 and Days 16-18 of a 28-day cycle in serial cohorts with doses of 750mg, 1000mg, 1250mg, 1500mg, 1750mg, and 2000mg.
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to see whether an altered schedule of giving erlotinib in combination with gemcitabine will be safe and might improve the results of the treatment for advanced cancer of the pancreas.

Gemcitabine and erlotinib are commercially available. Gemcitabine is FDA approved as first-line treatment for patients with locally advanced, unresectable or metastatic cancer of the pancreas. Erlotinib is FDA approved in combination with gemcitabine for the first-line treatment of patients with locally advanced, unresectable or metastatic pancreatic cancer.

The FDA recommended dose for erlotinib is 100 mg daily. This study will investigate the experimental administration of higher doses of erlotinib given for only three days twice a month, a schedule called "pulse dosing".

DETAILED DESCRIPTION:
Survival of pancreatic cancer patients remains poor, and treatment with erlotinib remains one of the few agents that have demonstrated increased survival. Alternative dosing schedules for erlotinib should be explored since chronic low dose therapy fails to achieve therapeutically effective concentrations for many patients and leads to increased skin toxicity and may induce acquired resistance without significantly impacting the tumor. Therefore, higher doses given for shorter periods of exposure, similar to the dosing of most chemotherapeutic agents, may achieve more effective therapeutic doses of than chronic low dose therapy and may minimize skin toxicity observed with erlotinib.

No phase I studies have been done with the combination of high dose pulse erlotinib therapy with gemcitabine. We propose a phase I dose escalation study of three day oral dosing of erlotinib with standard dose (1000 mg/m2) gemcitabine. The starting dose of erlotinib is 750 mg, approximately 50% of the the dose found to be safe in previous combination studies with carboplatin and paclitaxel and with pemetrexed [Riely et al. 2009, Davies et al. 2009]. Since acquired resistance can occur rapidly and 5 to 7 days of treatment is not better than 3 days of treatment, we will focus on a 3 day high-dose pulse treatment given every 14 days. This will provide 11 days between erlotinib dosing for the recovery of normal tissues. Levels of serum erlotinib will also be monitored due to considerable interpatient variability in the metabolism of erlotinib.

The hypotheses of this study are:

* High-dose pulse therapy with erlotinib can be safely administered with standard dose gemcitabine.
* High-dose pulse therapy with erlotinib will permit recovery of the epidermis between treatments resulting in reduced skin toxicity compared to chronic daily dosing.
* Disease control with high-dose pulse therapy may be superior to that with chronic low dose therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced pancreatic cancer defined as non-operable in a curative intent, locally recurrent, or metastatic disease.
* Measureable disease by (Response Evaluation Criteria in Solid Tumors) RECIST v1.1. Measureable lesions will be confirmed by radiological imaging.
* Progressive disease by (Response Evaluation Criteria in Solid Tumors) RECIST criteria during or after treatment with first-line chemotherapy (disease free interval must be less than 6 months) and have not received further second-line chemotherapy. Patients treated with prior chemo-radiation to the primary pancreatic tumor, for which the chemotherapeutic agent was used as a radio-sensitizing agent, are eligible.
* Age >18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0-2.
* Life expectancy of >2 months.
* Adequate laboratory parameters: All tests to be performed within 5 days prior to the first dose of erlotinib
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.
* Women of child bearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

* Radiation within 4 weeks of study enrollment. Radiotherapy not permitted while on study. Exception: palliative radiotherapy of metastasis in extremities is allowed, but such lesions cannot be used as target or non-target lesions.
* Investigational compound within 4 weeks of enrollment or who are planning to receive other investigational drugs while participating in the study.
* Chemotherapy, biologics, immunotherapy, vaccine, cytokine therapy within 4 weeks prior to enrollment.
* Presence of untreated and/or symptomatic central nervous system (CNS) metastasis.
* Severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months of study, chronic renal disease, chronic pulmonary disease or active uncontrolled infection).
* Known diagnosis of human immunodeficiency virus (HIV) infection.
* Presence of any other active or suspected acute or chronic uncontrolled infection or known symptomatic active hepatitis B or C.
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease.
* History of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer, cervical cancer in situ, localized biopsy-proven prostate cancer, or stage I colon cancer.
* Surgery within 3 weeks prior to enrollment.
* Patients taking Coumadin® or other agents containing warfarin, rivaroxaban, or dabigatran (exception: low dose Coumadin® (1 mg or less daily) administered prophylactically for maintenance of in-dwelling lines or ports is allowed).
* Patients taking any medications or substances that are inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A).
* Female patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities of each subject | 28 days
  Rate will be assessed through summaries of adverse events, clinical laboratory abnormalities, and changes in physical exam and vital signs. All subjects who receive a single dose of study medication will be considered evaluable for safety.

SECONDARY OUTCOMES:
Overall survival | 2 years
  the time from the first day of study treatment to date of death from any cause
progression-free survival | Up to 2 years
  the time from the first day of study treatment to date of disease progression
Best tumor response | up to 2 years
  a complete response (CR) or partial response (PR) as determined by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST)
Changes in the level of serum tumor marker cancer antigen (CA) 19-9 | up to 2 years
  changes evaluated via Fisher's exact tests or Wilcoxon rank sum tests, as appropriate
Adverse events related to pulse dose erlotinib and gemcitabine | From the initiation of study treatment and ends 30 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier
  description, timing, grade (Common Terminology Criteria for Adverse Events Version 4.03 [CTCAE v4.03]), severity, seriousness, and relatedness

CONTACTS AND LOCATIONS:
Overall Officials: Tony Reid, MD, PhD, Principal Investigator — University of California Medical Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States